CLINICAL TRIAL: NCT02494765
Title: Spatial Relationship of I-gelTM and Ambu® AuraOnceTM on Paediatric Airway: A Comparison on Three Dimensional MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mansoor Aqil, Associate Professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-14-1154
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Pediatric Laryngeal Mask Airway; Spatial Relations With Pediatric Airway; Assessed With Three Dimensional Magnetic Resonance Imaging
Keywords: I-gelTM; Ambu® AuraOnceTM; supraglottic devices; laryngeal mask effects on airway; 3D magnetic resonance imaging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I-gelTM (Active Comparator): I-gel is a supraglottic device made of gel like material. It is used for administration of anesthesia in selected patients.
  Interventions: Device: I-gel TM
- Ambu® AuraOnceTM (Active Comparator): Ambu AuraOnce (AO) is a supraglottic device having different material and its shaft has greater curvature than I-gel. It is also used for administration of anesthesia in selected patients.
  Interventions: Device: Ambu AuraOnce (AO)

INTERVENTIONS:
Device: I-gel TM — Airway management with I-gel
  Arms: I-gelTM
Device: Ambu AuraOnce (AO) — Airway management with Ambu AuraOnce (AO)
  Arms: Ambu® AuraOnceTM

SUMMARY:
At King Khalid University hospital approximately 1200-1500 MRI are done yearly on pediatric and neonatal patients. The investigating hospital is one of the pioneers in providing this service in the Kingdom (which was established about 10 years ago) to the patients of this age group. Only a small percentage of pediatric patients with age above 8 years accept the procedure to be done without anesthesia; and majority of MRI procedures are done under general anesthesia. The airway management of these patients is commonly accomplished with laryngeal mask airways (LMA).

LMA are in practice of anesthesia since early 1980s. Pediatric and neonatal patients (including ex-premature) have also been benefited by the use of LMA. There are many advantages of LMA over endotracheal tube (ETT) in pediatric patients like ease of insertion, securing airway rapidly, avoidance of muscle relaxants, reduced incidence of sore throat, post-operative hoarseness and coughing at the time of extubation, greater hemodynamic and intra ocular pressure (IOP) stability.

There are different types of pediatric LMAs available e.g. I-gel, ProSeal, LMA supreme, LMA classic, LMA unique, LarySeal and Ambu. These devices differ morphologically from each other (silicone, polyvinyl chloride or soft gel). Out of all this variety of LMAs only few are MRI compatible (do not produce any artifact in the MRI image), for example Ambu LMA and I-gel LMA and in King Khalid University Hospital (the investigating hospital) these two types are being used.

On search of literature the investigators found only one study in adults in which such comparison has been made and there was no study comparing different LMAs on the basis of their spatial effects on anatomical structures of the neck and airway in pediatric patients with age 12 years or below.

In this prospective randomized study, the investigators will compare the spatial relationship of I-gel Trademark (TM) and Ambu® AuraOnce (AO)TM on pediatric airway in pediatric patients undergoing 3-D MRI under general anesthesia (GA).

ELIGIBILITY:
Inclusion Criteria:

* After getting informed voluntary consent from the parents.
* American society of anesthesiologists (ASA) physical status I and II
* Age up to 12 years,
* Scheduled to undergo elective Magnetic resonance imaging (MRI) under General anesthesia (GA) for some medical or surgical disease of the -area (not involving oral cavity, larynx, pharynx and neck)
* Not likely to require use of muscle relaxants as MRI prerequisite (e.g breath holding).

Exclusion Criteria:

* Co-operative patients who will accept to undergo the procedure without anaesthesia
* Patients with upper respiratory tract infection, fever
* Known to be suffering from deformity of the face, larynx, pharynx or neck,
* Potentially difficult intubation,
* Full stomach patient,
* Contraindication to supraglottic device placement or GA,
* Failed supraglottic insertion or requiring emergency endotracheal intubation during the procedure -Patients whose trachea will already be intubated or will be having tracheostomy.-

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Effect on tongue | After 2 months
  The thickness of the tongue will be defined as the greatest distance between the surface of the tongue and the lower margin of the geniohyoideus muscle measured on sagittal T2 midline images. Scale (mm).

SECONDARY OUTCOMES:
Depth of intrusion of the tip of the supraglottic device into the Upper esophageal sphincter | After 2 months
  The depth of insertion relative to the glottis will be defined as the perpendicular distance between a horizontal line through the level of the glottis and a parallel line touching the tip of the supraglottic device on sagittal images. Scale (mm).
Effect of Supraglottic devices on hyoid bone | After 2months
  The position of the hyoid bone relative to cervical spine will be determined by measuring the shortest distance between the dorsal margin of the hyoid bone and the ventral margin of the opposing vertebra body. Scale (mm).
Effect of Supraglottic devices on glottic area | After 2 months
  The glottic area and the axial diagonal of the glottis will be measured on axial T1 slices at the narrowest part of the glottis after the images has been reoriented to be parallel to the vocal cords and the enclosed glottic area. Scale (mm).
Effect of Supraglottic devices on distance between common carotids | After 2 months
  The distance between the common carotids will be defined as the distance between the medial margins of the common carotid arteries measured on the same axial T1 section used to determine the glottic area. Scale (mm).
Effect of Supraglottic devices on the distance between the arytenoids | After 2 months
  The distance between the arytenoid cartilages will be measured on an axial T1 plane realigned as described above, with the points of measurement being the most medial part of the vocal process. Scale (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor Aqil, MD, Principal Investigator — King Saud University, King Khalid University hospital
Locations (1):
- King Saud University, King Khalid University Hospital, Riyadh, Saudi Arabia